CLINICAL TRIAL: NCT03799289
Title: Examination of the Feasibility and Preliminary Efficacy of Two Approaches for Improving Long-term Weight Loss
Brief Title: Approaches for Improving Long-term Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2096-18; R03DK115978-01A1 (NIH)
Record Dates: First submitted 2018-12-05; First posted 2019-01-10 (Actual); Results first posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-06

CONDITIONS: Obesity
Keywords: Obesity; Weight loss; physical activity; yoga; exercise
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iyengar Yoga (Experimental): Participants randomized to the yoga intervention arm will receive 12 weeks of group-based yoga instruction, following a 12-week standard behavioral weight loss program. Group-based yoga instruction will occur twice per week and classes will be 60 minutes in duration. The yoga program will consist of breathing, postural, and meditation practices and home-based yoga practice will also be prescribed.
  Interventions: Behavioral: Behavioral weight loss followed by yoga instruction
- Cooking/dietary education (Active Comparator): Participants randomized to the cooking/dietary education intervention arm will receive 12 weeks of group-based, cooking/dietary education instruction, following a 12-week standard behavioral weight loss program. This group-based instruction will occur twice per week and classes will be 60 minutes in duration. Classes will focus on providing basic nutrition knowledge and culinary skills, and will include cooking demonstrations.
  Interventions: Behavioral: Behavioral weight loss followed by cooking/dietary education instruction

INTERVENTIONS:
Behavioral: Behavioral weight loss followed by yoga instruction — 12-week standard behavioral weight loss program followed by a 12-week yoga intervention
  Arms: Iyengar Yoga
Behavioral: Behavioral weight loss followed by cooking/dietary education instruction — 12-week standard behavioral weight loss program followed by a 12-week cooking/dietary education intervention
  Arms: Cooking/dietary education

SUMMARY:
The purpose of this study is to examine two approaches for improving long-term weight loss success. All participants will receive a 12-week, in-person standard behavioral weight loss program followed by either 12 weeks of yoga instruction or 12 weeks of cooking/dietary education instruction (determined via randomization procedures). Assessments of weight, physical activity, dietary behaviors, and psychosocial factors will occur at baseline, 3, and 6 months.

DETAILED DESCRIPTION:
Behavioral weight loss (WL) programs result in clinically significant weight losses; however rates of long-term WL maintenance are poor. Previous studies suggest that long-term WL success may require an enhanced ability to overcome physiological and hedonic urges to eat and an improved capacity for dealing with life stressors, negative mood states, and food cravings. Thus interventions which target stress reduction and reduce the tendency to use food as a coping strategy for aversive experiences may offer a protective effect against dietary lapses; thereby improving long-term WL outcomes. Yoga is a mind-body intervention which reduces stress and improves overall physical and psychological well-being and offers promise for strengthening the psychological skill set needed for maintaining important weight-related behaviors long-term. The physical and cognitive skills practiced within yoga target multiple underlying psychological processes (e.g., mindfulness, distress tolerance) which could reduce emotional eating, improve dietary choices, and enhance one's ability to tolerate food cravings or hedonic urges to eat. While yoga is an effective treatment approach for other chronic health conditions, it has not been examined as a potential intervention for improving long-term WL outcomes. Within the context of the obesity field, yoga has been viewed as a mode of exercise and not necessarily as a mind-body intervention approach (as is the case in other fields). Thus, given the lower caloric expenditure of yoga in comparison to many forms of aerobic exercise, the effect of yoga on important weight- related processes and behaviors has not been examined.

The primary aims of this study are to examine the feasibility and acceptability of implementing yoga within a weight management program. Secondary aims focus on examining the impact of yoga, relative to a cooking/dietary education intervention (matched for contact time) on important psychological constructs (perceived stress, mindfulness, and distress tolerance) and weight. Sixty women with overweight or obesity will be randomly assigned to a 12-week standard behavioral WL program, followed by either 12 weeks of group-based yoga or 12 weeks of cooking/dietary information classes. Both groups will be instructed to self-monitor and achieve the dietary and aerobic exercise goals throughout the 24-week program. Primary assessments will occur at baseline and weeks 12 and 24.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-40 kg/m2
* Female

Exclusion Criteria:

* Presence of any condition that would limit one's ability to exercise or lose weight safely
* Recent weight loss
* Current or recent enrollment in a weight loss or mindfulness-based treatment program
* Women who are pregnant or planning on becoming pregnant
* History of a serious psychiatric disorder
* Recent cancer diagnosis (<1 year)
* Does not own a smartphone

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Unick, PhD, Principal Investigator — The Miriam Hospital's Weight Control & Diabetes Research Center
Locations (1):
- Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Initial Weight Loss Program (Weeks 1-12)
Arm/Group | Iyengar Yoga | Cooking/Dietary Education
Started | 30 | 30
Completed | 24 | 27
Not Completed | 6 | 3
Period: Maintenance Intervention (Weeks 13-24)
Arm/Group | Iyengar Yoga | Cooking/Dietary Education
Started | 24 | 27
Completed | 24 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 60 participants enrolled in this trial. A total of 51 completed the 12-week weight loss program and thus found out their randomization assignment to either the yoga or cooking/dietary education condition. Information presented is on those 51 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Iyengar Yoga | Cooking/Dietary Education | Total
Number analyzed (Participants) | 24 | 27 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (9.9) | 49.1 (9.5) | 48.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 27 | 51
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 20 | 25 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 19 | 23 | 42
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 27 | 51
Body mass index (BMI) at baseline (pre weight loss) [Mean (Standard Deviation); unit: kg /m^2] | 34.6 (4.1) | 34.5 (3.5) | 34.6 (3.8)
Body mass index (BMI) at 12 weeks (post weight loss intervention) [Mean (Standard Deviation); unit: kg/m^2] — Post-12 week weight loss was considered the 'new baseline' for those receiving the the yoga and cooking interventions, as we were examining these as intervention approaches for improving long-term weight loss
  kg/m^2 | 33.1 (4.5) | 31.8 (3.7) | 32.4 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Program Satisfaction Ratings
Description: Participants were asked, 'How satisfied were you with the yoga or cooking/dietary education intervention that you received over the past 3 months' on a 1-10 scale (1=very dissatisfied, 10=very satisfied)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Iyengar Yoga | Cooking/Dietary Education
Number analyzed (Participants) | 24 | 27
units on a scale | 7.6 (2.9) | 8.3 (2.4)

2. Primary Outcome: Intervention Session Attendance
Description: Yoga or control intervention sessions attended, expressed as a percentage (# of sessions completed/# of sessions possible x 100).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of sessions attended
Arm/Group | Iyengar Yoga | Cooking/Dietary Education
Number analyzed (Participants) | 24 | 27
percentage of sessions attended | 75.4 (24.6) | 75.9 (27.1)

3. Primary Outcome: Feasibility of the Intervention (Retention)
Description: Number of participants completing the 6-month assessment visit. Percentage of total participants can be computed as follows: the number of participants completing the 6-month assessment divided by the total number of participants who completed the 3-month weight loss program and learned of their randomization assignment
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Iyengar Yoga | Cooking/Dietary Education
Number analyzed (Participants) | 24 | 27
Participants | 24 | 27

4. Secondary Outcome: Changes in Perceived Stress (Measured Via the Perceived Stress Scale)
Description: Perceived stress scores range from 0-40, with higher scores indicating higher perceived stress. Change in perceived stress was calculated as follows: 24-week perceived stress score minus 12-week perceived stress score. Negative change scores indicate that perceived stress was reduced as a result of the yoga or cooking/dietary education intervention whereas positive scores indicate that perceived stress increased.
Time Frame: Change from 12 to 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Iyengar Yoga | Cooking/Dietary Education
Number analyzed (Participants) | 24 | 27
units on a scale | 0.01 (0.51) | -0.06 (0.60)

5. Secondary Outcome: Change in Dispositional Mindfulness (Assessed Via the Five Facet Mindfulness Questionnaire) - Observing Subscale
Description: The observation subscale assesses the ways we use our sensory awareness. It involves how we see, feel, and perceive the internal and external world around us and select the stimuli that require our attention and focus. Mindfulness subscale scores range from 8-40, with higher scores indicating greater mindfulness. Change in mindfulness subscale was calculated as follows: 24-week mindfulness subscale score minus 12-week mindfulness subscale score. Negative change scores indicate that mindfulness was reduced as a result of the yoga or cooking/dietary education intervention whereas positive scores indicate that mindfulness increased.
Time Frame: Change from 12 to 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Iyengar Yoga | Cooking/Dietary Education
Number analyzed (Participants) | 24 | 27
units on a scale | 1.7 (5.9) | 0.9 (3.7)

6. Secondary Outcome: Change in Dispositional Mindfulness (Assessed Via the Five Facet Mindfulness Questionnaire) - Describing Subscale
Description: The describing subscale evaluates the way we label our experiences and express them in words to ourselves and others. Subscale scores range from 8-40, with higher scores indicating greater mindfulness. Change in mindfulness subscale was calculated as follows: 24-week mindfulness subscale score minus 12-week mindfulness subscale score. Negative change scores indicate that mindfulness was reduced as a result of the yoga or cooking/dietary education intervention whereas positive scores indicate that mindfulness increased.
Time Frame: Change from 12 to 24 weeks
Measure: Mean (Standard Deviation); unit: Change on a scale
Arm/Group | Iyengar Yoga | Cooking/Dietary Education
Number analyzed (Participants) | 24 | 27
Change on a scale | -0.17 (5.1) | -0.9 (3.9)

7. Secondary Outcome: Change in Dispositional Mindfulness (Assessed Via the Five Facet Mindfulness Questionnaire) - Acting With Awareness Subscale
Description: This subscale examines whether we can act out of quick judgment and get out of the autopilot mode before responding to a situation. Subscale scores range from 8-40, with higher scores indicating greater mindfulness. Change in mindfulness subscale was calculated as follows: 24-week mindfulness subscale score minus 12-week mindfulness subscale score. Negative change scores indicate that mindfulness was reduced as a result of the yoga or cooking/dietary education intervention whereas positive scores indicate that mindfulness increased.
Time Frame: Change from 12 to 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Iyengar Yoga | Cooking/Dietary Education
Number analyzed (Participants) | 24 | 27
units on a scale | -0.29 (3.06) | 0.04 (5.03)

8. Secondary Outcome: Change in Dispositional Mindfulness (Assessed Via the Five Facet Mindfulness Questionnaire) - Non-judgmental Inner Critic Subscale
Description: This subscale assesses the degree of self-acceptance and unconditional empathy for oneself and others. Subscale scores range from 8-40, with higher scores indicating greater mindfulness. Change in mindfulness subscale was calculated as follows: 24-week mindfulness subscale score minus 12-week mindfulness subscale score. Negative change scores indicate that mindfulness was reduced as a result of the yoga or cooking/dietary education intervention whereas positive scores indicate that mindfulness increased.
Time Frame: Change from 12 to 24 weeks
Measure: Mean (Standard Deviation); unit: Change on a scale
Arm/Group | Iyengar Yoga | Cooking/Dietary Education
Number analyzed (Participants) | 24 | 27
Change on a scale | 0.46 (4.34) | 0.74 (4.59)

9. Secondary Outcome: Change in Dispositional Mindfulness (Assessed Via the Five Facet Mindfulness Questionnaire) - Non-reactivity Subscale
Description: This subscale assesses active detachment from negative thoughts and emotions so that we can accept their existence and choose not to react to them. Subscale scores range from 7-35, with higher scores indicating greater mindfulness. Change in mindfulness subscale was calculated as follows: 24-week mindfulness subscale score minus 12-week mindfulness subscale score. Negative change scores indicate that mindfulness was reduced as a result of the yoga or cooking/dietary education intervention whereas positive scores indicate that mindfulness increased.
Time Frame: Change from 12 to 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Iyengar Yoga | Cooking/Dietary Education
Number analyzed (Participants) | 24 | 27
units on a scale | 0.33 (3.17) | -1.67 (3.82)

10. Secondary Outcome: Change in Distress Tolerance (Assessed Via the Distress Tolerance Scale)
Description: The Distress Tolerance Scale is a 15-item measure designed to assess one's perceived ability to tolerate emotional distress. Total scores range from 15-75 with higher scores on the scale indicate greater levels of distress tolerance. Change in distress tolerance was calculated as follows: 24-week distress tolerance score minus 12-week distress tolerance score. Negative change scores indicate that distress tolerance decreased as a result of the yoga or cooking/dietary education intervention whereas positive scores indicate that distress tolerance increased.
Time Frame: Change from 12 to 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Iyengar Yoga | Cooking/Dietary Education
Number analyzed (Participants) | 24 | 27
units on a scale | 0.02 (0.51) | -0.06 (0.60)

11. Secondary Outcome: Change in Weight
Description: Calculated as the percentage of weight lost from 12 to 24 weeks, as a result of the yoga or cooking/dietary education interventions. It was calculated as follows: (24-week weight minus 12-week weight) / 12-week weight x 100. Positive numbers indicate weight gain whereas negative numbers indicate weight loss.
Time Frame: Change from 12 to 24 weeks
Measure: Mean (Standard Deviation); unit: Percent weight change
Arm/Group | Iyengar Yoga | Cooking/Dietary Education
Number analyzed (Participants) | 24 | 27
Percent weight change | -0.33 (2.91) | -0.38 (4.03)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Iyengar Yoga | Cooking/Dietary Education
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/27
Other Adverse Events (participants affected / at risk) | 0/24 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT03799289/Prot_SAP_002.pdf
  • Informed Consent Form (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/89/NCT03799289/ICF_000.pdf